CLINICAL TRIAL: NCT04725370
Title: Comparison of Cleft Lip and Palate Between a United States Tertiary Care Center and a Guatemalan Surgical Mission: A Cohort Study of 629 Pediatric Patients and a Survey of Risk Factors
Brief Title: Characterization of Cleft Lip and Palate Conditions in Guatemala
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 19-016144
Record Dates: First submitted 2021-01-04; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cleft Lip; Cleft Palate; Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CHOP (US): Children with isolated cleft lip and/or cleft palate scheduled for surgery between 2012 to 2019 at the Children's Hospital of Philadelphia, Philadelphia, PA, USA.
- SFG (Guatemala): Children with isolated cleft lip and/or cleft palate scheduled for surgery between 2017 and 2020 with Smiles for Guatemala, Guatemala City, Guatemala.
  Interventions: Other: NA - survey instrument

INTERVENTIONS:
Other: NA - survey instrument — Survey instrument was administered verbally to parents of the Guatemalan cohort.
  Groups: SFG (Guatemala)

SUMMARY:
The purpose of this study is to compare types of and risk factors for cleft lip and palate in a Guatemalan population to a United States population.

DETAILED DESCRIPTION:
Demographic, surgical, and cleft type data from US patients were gathered via chart review of the electronic medical record. Data from Guatemalan patients was gathered orally from patient caregivers in their native language. Consent was also given orally in the caregivers native language. All data was de-identified prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of isolated cleft lip and/or palate
* scheduled for cleft-related surgery at either the Children's Hospital of Philadelphia or Smiles for Guatemala during the previously described time frames

Exclusion Criteria:

* diagnosis of a recognized medical syndrome
* medically complex defined as having major medical problems in three or more organ systems
* diagnosis of isolated midline cleft lip
* diagnosis of Tessier facial cleft
* greater than 18 years of age

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with isolated cleft lip and/or palate scheduled for cleft-related surgery at either the Children's Hospital of Philadelphia or Smiles for Guatemala during the previously described time frames
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Cleft phenotype | pre-surgery
  Presence, laterality, and completeness of cleft lip and/or palate as classified by the LAHSHAL system, data gathered by physical exam

SECONDARY OUTCOMES:
Cleft risk factors | during the surgery
  Presence of potential risk factors for cleft lip and palate such as maternal exposures during pregnancy, data gathered by interview with caregivers
Surgical care | pre-surgery
  Type of surgery scheduled and patient age at time of scheduled surgery, data gathered by chart review

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A Jackson, MD, Principal Investigator — Children's Hospital of Philadelphia; Michelle Scott, DDS, MBA, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided